CLINICAL TRIAL: NCT03509129
Title: Evaluating Columbia Moves: A Social Network Approach Using a Team Competition and Technology to Increase Physical Activity
Brief Title: Columbia Moves Physical Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018
Record Dates: First submitted 2018-04-16; First posted 2018-04-26 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-04

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — PLEKHG5 protein, human; Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TECH (Technology) (Active Comparator): Participants will receive a theory-based physical activity program. They will enroll in the study as part of a self-selected group of 3-8 individuals. They will be provided with a personal step goal and Fitbit Alta HR for self-monitoring physical activity. They will also have access to a study website that will be accessible across conventional and mobile platforms. They will be asked to visit the website each week to receive behavior change information and guidance.
  Interventions: Behavioral: TECH (Technology)
- TECH+COMP (Technology + Competition) (Experimental): Participants will receive the same intervention components as the TECH goup, as well as a study designed team competition.
  Interventions: Behavioral: TECH+COMP (Technology + Competition)

INTERVENTIONS:
Behavioral: TECH (Technology) — Participants will receive a theory-based physical activity program. They will enroll in the study as part of a self-selected group of 3-8 individuals. They will be provided with a personal step goal and Fitbit Alta HR for self-monitoring physical activity. They will also have access to a study website that will be accessible across conventional and mobile platforms. They will be asked to visit the website each week to receive behavior change information and guidance.
  Device: Fitbit Alta HR
  Arms: TECH (Technology)
Behavioral: TECH+COMP (Technology + Competition) — Participants will receive the same intervention components as the TECH group, as well as a team competition. The competition will be based on the following two aspects: total daily steps accumulated relative to group size and total number of points retained for achieving weekly physical activity challenges.
  Device: Fitbit Alta HR
  Arms: TECH+COMP (Technology + Competition)

SUMMARY:
The purpose of this study is to evaluate the effect of adding a team competition comprised of members of existing social networks to a technology-delivered program for enhancing physical activity among insufficiently active adults.

DETAILED DESCRIPTION:
This 3-month randomized controlled trial is designed to investigate the efficacy and feasibility of a novel, technology-oriented physical activity intervention characterized by existing social networks and a team competition. Participants will be recruited via emails, fliers, and word of mouth. They will be randomized to a technology-mediated physical activity treatment (TECH) or a treatment which receives an identical intervention as TECH plus a study designed team competition for physical activity promotion (TECH+COMP).

ELIGIBILITY:
Inclusion Criteria:

* Insufficiently active as determined by a one-week, accelerometer-based physical activity measurement
* Body mass index (BMI) between 25 kg/m2 and 55 kg/m2
* Between ages 18 and 65 years
* Access to computer with Internet connection
* Smartphone ownership (Android or iOS)
* Willing to be randomized to either one of the two study groups
* Part of a self-selected team of 3-8 eligible individuals
* Members of the same household cannot be part of separate groups
* Able to walk at least 1/4 mile without stopping

Exclusion Criteria:

* Currently lactating, pregnant, or planning to become pregnant during the length of the study
* Diagnosed with type 1 or type 2 diabetes
* Medical or physical contraindications or limitations for engaging in physical activity
* History of major medical or psychiatric conditions
* Currently participating in a physical activity program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Accelerometer-measured change from Baseline Daily Steps at 3 months and 12 months | 0, 3, and 12 months
  Change in daily steps

SECONDARY OUTCOMES:
Accelerometer-measured change from Baseline Minutes of Moderate-to-Vigorous Physical Activity at 3 months and 12 months | 0, 3, and 12 months
  Change in moderate-to-vigorous physical activity
Change from Baseline in Perceived Social Support for Exercise (Sallis Social Support and Exercise Survey) at 3 and 12 months | 0, 3, and 12 months
  Change in perceived social support for exercise (scale total score range: 1 to 5, with 1 representing low perceived social support for exercise and 5 representing high perceived social support for exercise; responses to all items are averaged to yield a total final score)

OTHER OUTCOMES:
Participant Satisfaction (Satisfaction Questionnaire) | 4 months
  Participant satisfaction with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Monroe, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Data will only be reported in aggregate.

REFERENCES:
- [Derived] Monroe CM, Cai B, Edney S, Jake-Schoffman DE, Brazendale K, Bucko A, Armstrong B, Yang CH, Turner-McGrievy G. Harnessing technology and gamification to increase adult physical activity: a cluster randomized controlled trial of the Columbia Moves pilot. Int J Behav Nutr Phys Act. 2023 Nov 3;20(1):129. doi: 10.1186/s12966-023-01530-1. PMID 37924083